CLINICAL TRIAL: NCT03878277
Title: Coffee, Renal Oxygenation, Blood Flow and Glomerular Filtration Rate in Early Diabetic Kidney Disease.
Brief Title: Evaluation of Coffee Therapy for Improvement of Renal Oxygenation
Acronym: COFFEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-1874
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Type1diabetes; Type1 Diabetes Mellitus; Diabetic Kidney Disease; Juvenile Diabetes; Diabetic Nephropathies; Diabetes Complications; Diabetes, Autoimmune
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 1; Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cold Brew Coffee (Experimental): 6 days of drinking 1 bottle of Starbucks® Cold brew 325ml [205 mg caffeine] every morning between 6am-9am.
  Interventions: Drug: Starbucks® Cold brew - 325ml bottle

INTERVENTIONS:
Drug: Starbucks® Cold brew - 325ml bottle — Starbucks® Cold brew 325ml bottles daily [205mg caffeine] will be provided to the participants. Participants will be instructed to drink 1 bottle every morning between 6 and 9 am for 6 days prior to the post-intervention visit. The 7th day is the post-intervention visit, and participants will be asked to drink 1 bottle the morning of the study visit

SUMMARY:
Over 1.25 million Americans have Type 1 Diabetes (T1D), increasing risk for early death from cardiovascular disease (CVD). Despite advances in glycemic and blood pressure control, a child diagnosed with T1D is expected to live up to 17 years less than non-diabetic peers. The strongest risk factor for CVD and mortality in T1D is diabetic kidney disease (DKD). Current treatments, such as control of hyperglycemia and hypertension, are beneficial, but only partially protect against DKD. This limited progress may relate to a narrow focus on clinical manifestations of disease, rather than on the initial metabolic derangements underlying the initiation of DKD. Renal hypoxia, stemming from a potential metabolic mismatch between increased renal energy expenditure and impaired substrate utilization, is increasingly proposed as a unifying early pathway in the development of DKD. T1D is impacted by several mechanisms which increase renal adenosine triphosphate (ATP) consumption and decrease ATP generation.

Caffeine, a methylxanthine, is known to alter kidney function by several mechanisms including natriuresis, hemodynamics and renin-angiotensin-aldosterone system. In contrast, to other natriuretic agents, caffeine is thought to fully inhibit the local tubuloglomerular feedback (TGF) response to increased distal sodium delivery. This observation has broad-ranging implications as caffeine can reduce renal oxygen (O2) consumption without impairing effective renal plasma flow (ERPF) and glomerular filtration rate (GFR).

There are also data suggesting that chemicals in coffee besides caffeine may provide important cardio-renal protection. Yet, there are no data examining the impact of coffee-induced natriuresis on intrarenal hemodynamic function and renal energetics in youth-onset T1D. Our overarching hypothesis in the proposed pilot and feasibility trial is that coffee drinking improves renal oxygenation by reducing renal O2 consumption without impairing GFR and ERPF. To address these hypotheses, we will measure GFR, ERPF, renal perfusion and oxygenation in response to 7 days of cold brew coffee (one Starbucks® Cold brew 325ml bottle daily [205mg caffeine]) in an open-label pilot and feasibility trial in 10 adolescents with T1D already enrolled in the CASPER Study (PI: Bjornstad).

ELIGIBILITY:
Inclusion Criteria:

* Youth with T1D (antibody +) with <10 year duration
* Age 12-21 years
* Weight >57 lbs and <350 lbs
* BMI >5th %ile
* HbA1c <12%
* Previous exposure to caffeine

Exclusion Criteria:

* Anemia
* Allergy to shellfish or iodine
* Severe illness, recent diabetic ketoacidosis (DKA)
* Tachyarrhythmias, Attention-deficit/hyperactivity disorder (ADHD), tremors, tics, Tourette's, arrythmias, insomnia, overactive bladder
* Estimated Glomerular Filtration Rate (eGFR) <60 ml/min/1.73 m2 or creatinine > 1.5 mg/dl or history of albumin-to-creatinine ratio (ACR) >300 mg/g
* MRI Scanning contraindications (claustrophobia, implantable metal devices that are non-MRI compatible, >350 lbs)
* Pregnancy or nursing
* (Angiotensin-converting enzyme) ACE inhibitors, angiotensin receptor blockers (ARBs), diuretics, sodium-glucose co-transport (SGLT) 2 or 1 blockers, daily NSAIDs or aspirin, sulfonamides, thiazolsulfone or probenecid, atypical antipsychotics, steroids

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petter Bjornstad, MD, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cold Brew Coffee
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cold Brew Coffee
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.5 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 10

OUTCOME MEASURES:

1. Primary Outcome: Renal Oxygenation
Description: Measured by blood oxygen level dependent (BOLD MRI), before and after Lasix injection;Regions of interest (ROI) analysis for BOLD MRI will be performed on a Leonardo Workstation (Siemens Medical Systems, Germany). Typically, 1 to 3 regions in each, cortex and medulla, per kidney per slice will be defined leading to a total of about 10 ROIs per region (cortex and medulla) per subject. The mean and standard deviation of these 10 measurements will be used a R2* measurement for the region, for the subject and for that time point. Additionally, two (delta) R2*s will be calculated as defined below:
  (delta) R2*(medulla, furosemide) = R2* (medulla, pre-furosemide) - R2* (medulla, post-furosemide); (delta) R2*(cortex, medulla) = Baseline R2* (medulla) - Baseline R2* (cortex).
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Cold Brew Coffee
Number analyzed (Participants) | 10
s^-1
  Before cold brew | 22.4 (1.5)
  After cold brew | 22.5 (2.1)

2. Primary Outcome: Renal Perfusion
Description: Measured by pseudocontinuous arterial spin labeling (pCASL) MRI; ROI analysis will be used to estimate (delta) M (difference in signal intensity between non-selective and selective inversion images). Using the same ROI, M0 will be estimated from the proton density image. T1 measurements from the same ROI will be obtained by fitting the signal intensity vs. inversion time data as described previously (104) using XLFit (ID Business Solutions Ltd., UK) or T1 maps created using MRI Mapper (Beth Israel Deaconess Medical Center, Boston). Partition coefficient will be assumed to be 0.8 ml/gm (105, 106). These values will then be used to estimate regional blood flow.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: ml/s/100g
Arm/Group | Cold Brew Coffee
Number analyzed (Participants) | 10
ml/s/100g
  Before cold brew (Right kidney ASL) | 3.02 (0.67)
  After cold brew (Right kidney ASL) | 3.03 (0.62)
  Before cold brew (Left kidney ASL) | 3.15 (0.50)
  After cold brew (Left kidney ASL) | 3.03 (0.72)

3. Secondary Outcome: Glomerular Filtration Rate
Description: Measured by Iohexol clearance; An intravenous (IV) line was placed, and participants were asked to empty their bladders. Spot plasma and urine samples were collected prior to iohexol infusion. Iohexol was administered through bolus IV injection (5 mL of 300 mg/mL; Omnipaque 300, GE Healthcare). An equilibration period of 120 min was used and blood collections for iohexol plasma disappearance were drawn at +120, +150, +180, +210, +240 min (11). Because the Brøchner-Mortensen equation underestimates high values of GFR, the Jødal-Brøchner-Mortensen equation was used to calculate the GFR (12). We report absolute GFR (mL/min) and RPF (mL/min) in the main analyses because the practice of indexing GFR and RPF for body surface underestimates hyperfiltration and hyperperfusion (14), and body surface area (BSA) calculations introduce noise into the clearance measurements.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Cold Brew Coffee
Number analyzed (Participants) | 10
ml/s
  Before cold brew | 3.25 (0.47)
  After cold brew | 3.27 (0.80)

4. Secondary Outcome: Effective Renal Plasma Flow
Description: Measured by para-aminohippurate (PAH) clearance; An intravenous (IV) line was placed, and participants were asked to empty their bladders. Spot plasma and urine samples were collected prior PAH infusion. PAH (2 g/10 mL, prepared at the University of Minnesota, with a dose of [weight in kg]/75 × 4.2 mL; IND #140129) was given slowly over 5 min followed by a continuous infusion of 8 mL of PAH and 42 mL of normal saline at a rate of 24 mL/h for 2 h. After an equilibration period, blood was drawn at 90 and 120 min, and RPF was calculated as PAH clearance divided by the estimated extraction ratio of PAH, which varies by the level of GFR (13). We report absolute GFR (mL/min) and RPF (mL/min) in the main analyses because the practice of indexing GFR and RPF for body surface underestimates hyperfiltration and hyperperfusion (14), and body surface area (BSA) calculations introduce noise into the clearance measurements.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Cold Brew Coffee
Number analyzed (Participants) | 10
ml/s
  Before cold brew | 13.08 (1.58)
  After cold brew | 13.02 (0.67)

5. Secondary Outcome: Tubular Injury Markers
Description: Measured by markers of kidney injury in plasma; Cystatin C (mg/L) was measured by immunoturbidimetric method (Kamiya Biomedical) by our Clinical Translational Research Center Core Laboratory.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cold Brew Coffee
Number analyzed (Participants) | 10
mg/L
  Before cold brew (cystatin C) | 0.82 (0.18)
  After cold brew (cystatin C) | 0.84 (0.19)

ADVERSE EVENTS:
Time Frame: During the duration of trial with cold brew (7 days) as well as 24 hours after the last study visit.
Arm/Group | Cold Brew Coffee
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cold Brew Coffee (N=10)
Vasovagal syncope (Vascular disorders) | 1 — Participant reported experiencing dizziness and lightheadedness during manipulation of peripheral IV by nursing staff during the hyperglycemic clamp. Participant given option to leave or continue in study. Participant chose to finish the study visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT03878277/Prot_SAP_000.pdf